CLINICAL TRIAL: NCT00589849
Title: T-Wave Alternans in Acute Myocardial Infarction: An Evaluation of the Time of Testing on Its Prognostic Accuracy
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 05-13651; 05-13651
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Results first posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-09

CONDITIONS: Myocardial Infarction; Arrhythmias
Keywords: Myocardial Infarction; Arrhythmia; T-wave alternans
MeSH Terms: conditions — Myocardial Infarction; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: T-wave Alternans

INTERVENTIONS:
Procedure: T-wave Alternans — T-wave alternans is an electrocardiographic finding that is defined as the beat-to beat fluctuation in the amplitude or shape of T wave

SUMMARY:
T-wave alternans is an electrocardiographic finding that has been shown to predict the occurrence of future cardiac arrhythmias in patients who have had a heart attack. What is unknown about T-wave alternans testing is when is the best time to perform the test. In most studies, T-wave alternans testing is conducted 4 weeks or more after a heart attack. It is unknown if T-wave alternans testing performed prior to hospital discharge in heart attack patients is reliable. The objective of this project is to determine the diagnostic accuracy of T-wave alternans testing performed prior to hospital discharge and again at 30 days after hospital discharge in patients who have suffered a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myocardial Infarction (MI) confirmed by electrocardiographic and or/ enzymatic criteria
* Patients with a left ventricular ejection fraction of 45% or less

Exclusion Criteria:

* Patients with (1) atrial fibrillation, (2) pacemaker rhythm, (3) left bundle branch block, (4) class III-IV heart failure, (5) inability to achieve a target heart rate with exercise or handgrip stress or (6) spontaneous sustained ventricular tachycardia/ventricular fibrillation will be excluded
* Patients with recurrent angina pectoris, MI, coronary revascularization, or any other adverse cardiovascular event in the 30 days following their initial MI will also be excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aryan Mooss, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T Wave Altenans Stress Test
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | T Wave Altenans Stress Test
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Diagnostic Accuracy of TWA in Predicting Arrhythmic Events, Cardiovascular Mortality, and Total Mortality in Patients With Acute MI
Time Frame: 30 days
Reporting Status: Not Posted

2. Primary Outcome: Event Free Survival at 1 Year
Description: Survival without ventricular tachycardia/ventricular fibrillation (VT/VF) or sudden cardiac death at 1 year
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | T Wave Altenans Stress Test
Number analyzed (Participants) | 32
participants | 32

ADVERSE EVENTS:
Arm/Group | T Wave Altenans Stress Test
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes